CLINICAL TRIAL: NCT04099030
Title: The Effects of the Opioid Drug Shortages on Selection of Nonopioid Analgesics During Laparoscopic Cholecystectomy
Brief Title: Effect of Opioid Shortage on Drug Selection
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00057062
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2019-09

CONDITIONS: Opioid Use, Unspecified
Keywords: drug shortage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Opioid shortage: Patients undergoing laparoscopic cholecystectomy during time of Fentanyl drug shortage
- Normal Opioid supply (no shortage): Patients undergoing laparoscopic cholecystectomy during time of normal Fentanyl drug supply

SUMMARY:
This study will look at the effects of fentanyl shortage in laparoscopic cholecystectomy cases. The opioid shortage, specifically hydromorphone and fentanyl, caused a decrease in administration of opioid analgesia for laparoscopic cholecystectomy intraoperatively.

DETAILED DESCRIPTION:
The goal of this study is to look at the clinical impact of the drug shortage of intravenous (IV) opioids from 2016 to 2018. IV opioids are used in the hospital setting ranging from the Emergency Department to the Intensive Care Unit (ICU) to the Operating room. This study will look at the usage of IV opioids in the operating room setting and determine how practice has change in the setting of drug shortage. The study team hypothesizes that the average monthly consumption of fentanyl and hydrophone would have been decreased for laparoscopic cholecystectomy intraoperatively during the opioid shortage period as compared to before the shortage period.

ELIGIBILITY:
Inclusion Criteria:

* All Genders
* History of laparoscopic cholecystectomy
* American Society of Anesthesiologist classification (ASA) 1-4 emergent and Non emergent
* Adult >18 years old
* Wake Forest Baptist Medical Center Main Operating rooms

Exclusion Criteria:

* Regional Anesthetic
* ASA 5 and 6

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Laparoscopic Cholecystectomy at Wake Forest Baptist Medical Center General ORS
Sampling Method: Non-Probability Sample
Enrollment: 1668 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Total Fentanyl usage | September 2016 to August 2017
  Monthly average amount administered per case per kg
Total Fentanyl usage | September 2017 to May 2018
  Monthly average amount administered per case per kg
Total Fentanyl usage | June 2018 to May 2019
  Monthly average amount administered per case per kg

SECONDARY OUTCOMES:
Nonopioid analgesia usage | September 2016 to August 2017
  Monthly average amount administered per case per kg
Nonopioid analgesia usage | September 2017 to May 2018
  Monthly average amount administered per case per kg
Nonopioid analgesia usage | June 2018 to May 2019
  Monthly average amount administered per case per kg
Number of CPR incidents | September 2016 to August 2017
  post-operative complication
Number of CPR incidents | September 2017 to May 2018
  post-operative complication
Number of CPR incidents | June 2018 to May 2019
  post-operative complication
Number of reintubation incidents | September 2016 to August 2017
  post-operative complication
Number of reintubation incidents | September 2017 to May 2018
  post-operative complication
Number of reintubation incidents | June 2018 to May 2019
  post-operative complication
Number of incidents requiring administration of emergency drugs | September 2016 to August 2017
  post-operative complication
Number of incidents requiring administration of emergency drugs | September 2016 to May 2018
  post-operative complication
Number of incidents requiring administration of emergency drugs | June 2018 to May 2019
  post-operative complication
Length of hospital stay | September 2016 to August 2017
Length of hospital stay | September 2016 to May 2018
Length of hospital stay | June 2018 to May 2019

OTHER OUTCOMES:
Postoperative Pain Scores | September 2016 to August 2017
  Pain scores range from 0 to 10 with higher score denoting more pain
Postoperative Pain Scores | September 2017 to May 2018
  Pain scores range from 0 to 10 with higher score denoting more pain
Postoperative Pain Scores | June 2018 to May 2019
  Pain scores range from 0 to 10 with higher score denoting more pain
Time Spent in Post-anesthesia Care Unit (PACU) | September 2016 to August 2017
Time Spent in Post-anesthesia Care Unit (PACU) | September 2017 to May 2018
Time Spent in Post-anesthesia Care Unit (PACU) | June 2018 to May 2019

CONTACTS AND LOCATIONS:
Overall Officials: Scott Miller, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klaus DA, de Bettignies AM, Seemann R, Krenn CG, Roth GA. Impact of a remifentanil supply shortage on mechanical ventilation in a tertiary care hospital: a retrospective comparison. Crit Care. 2018 Oct 26;22(1):267. doi: 10.1186/s13054-018-2198-3. PMID 30367645